CLINICAL TRIAL: NCT03233139
Title: A Phase 1 Study to Investigate the Safety and Pharmacokinetics of Cemiplimab (Anti-PD-1) and Other Agents in Japanese Patients With Advanced Malignancies
Brief Title: Safety and Pharmacokinetics of Cemiplimab Anti-programmed Death-ligand 1 (Anti-PD-1) and Other Agents in Japanese Adult Patients With Advanced Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1622
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Advanced Malignancies
Keywords: Japanese patients
MeSH Terms: interventions — cemiplimab; Ipilimumab; Gemcitabine; Pemetrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Cemiplimab (Experimental): Part 1
  Interventions: Drug: Cemiplimab
- Cohort A (Experimental): Part 2
  Interventions: Drug: Cemiplimab
- Cohort B (Experimental): Part 2
  Interventions: Drug: Cemiplimab; Drug: Ipilimumab; Drug: Platinum-doublet chemotherapy; Drug: Gemcitabine; Drug: Pemetrexed; Drug: Paclitaxel
- Cohort C (Experimental): Part 2
  Interventions: Drug: Cemiplimab; Drug: Platinum-doublet chemotherapy; Drug: Pemetrexed; Drug: Paclitaxel
- Cohort D (Experimental): Part 2
  Interventions: Drug: Cemiplimab; Drug: Fianlimab
- Cohort E (Experimental): Part 2
  Interventions: Drug: Cemiplimab; Drug: Platinum-doublet chemotherapy; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Fianlimab

INTERVENTIONS:
Drug: Cemiplimab — Patients will be administered cemiplimab as per protocol. For Cohort A Only, patients with confirmed progressive disease may opt to receive up to 4 cycles of platinum doublet chemotherapy in addition to cemiplimab per investigator's judgement.
  Other Names: REGN2810; Libtayo
Drug: Ipilimumab — To be administered per protocol
  Arms: Cohort B
Drug: Platinum-doublet chemotherapy — To be administered per protocol
  Arms: Cohort B; Cohort C; Cohort E
Drug: Gemcitabine — To be administered per protocol
  Other Names: Gemzar
  Arms: Cohort B
Drug: Pemetrexed — To be administered per protocol
  Other Names: Alimta
  Arms: Cohort B; Cohort C; Cohort E
Drug: Paclitaxel — To be administered per protocol
  Other Names: Taxol
  Arms: Cohort B; Cohort C; Cohort E
Drug: Fianlimab — To be administered per protocol
  Arms: Cohort D; Cohort E

SUMMARY:
Part 2 Cohorts A and C This study is being conducted to test the safety and pharmacokinetics of cemiplimab in patients with lung cancer. The study is also being conducted to test if cemiplimab, alone or in combination, can reduce the size of your tumor by helping the immune system destroy the tumor.

Part 2 Cohorts D and E This study is being conducted to test the safety and pharmacokinetics of fianlimab and cemiplimab in patients with lung cancer. The study is also being conducted to test if fianlimab and cemiplimab, with or without chemotherapy, can reduce the size of your tumor by helping the immune system destroy the tumor.

ELIGIBILITY:
Key Inclusion Criteria:

1. Disease types under study:

   * Part 1: Histologically or cytologically confirmed diagnosis of malignancy with no alternative standard-of-care therapeutic option
   * Part 2: Patients with histologically or cytologically documented squamous or non-squamous NSCLC with stage IIIB or IIIC or stage IV disease who received no prior systemic treatment for recurrent or metastatic NSCLC.
   * Patients in Part 2 NSCLC cohorts must have available archival or newly obtained formalin-fixed tumor tissue from a metastatic/recurrent site, which has not previously been irradiated.
2. ECOG (Eastern Cooperative Oncology Group) PS (Performance status) ≤1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature [eg, light housework or office work]). Note: Patients with ECOG PS >1 are ineligible.
3. Patients must have been born in Japan, and their biological parents and grandparents must all have been of Japanese origin
4. Willing and able to comply with clinic visits and study-related procedures
5. For Part 2, Cohorts D and E: Available tissue for retrospective testing using assay performed by a central laboratory, as specified in the study manual.

Key Exclusion Criteria:

1. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that requires treatment with systemic immunosuppressive treatments, which may suggest risk for Immune-mediated adverse event (imAE)s. The following are not exclusionary: vitiligo, childhood asthma that has resolved, residual hypothyroidism that requires only hormone replacement or psoriasis that does not require systemic treatment.
2. Untreated brain metastasis (es) that may be considered active. Patients with previously treated brain metastases may participate provided they are stable, there is no evidence of new or enlarging brain metastases, and the patient does not require any systemic corticosteroids for management of brain metastases within 4 weeks prior to the first dose of cemiplimab.
3. Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of cemiplimab.
4. Any positive test (ribonucleic acid (RNA) or Deoxyribonucleic acid (DNA) by polymerase chain reaction) for hepatitis B, hepatitis C, or human immunodeficiency virus indicating uncontrolled active or chronic infection.
5. History of pneumonitis or interstitial lung disease
6. Surgery within 1 month of first dose and radiation therapy within 2 weeks of first dose
7. Completed palliative radiation therapy within the prior 2 weeks or has not recovered from any medically significant radiation-related Adverse Event (AE)
8. Patients that have never smoked, defined as smoking ≤100 cigarettes in a lifetime (Part 2)
9. Patients with tumors tested positive for epidermal growth factor receptor (EGFR) gene mutations, anaplastic lymphoma kinase (ALK) gene translocations, or ROS1 fusions (Part 2)

Note: Other protocol defined inclusion/exclusion criteria apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) in patients treated with cemiplimab as monotherapy | Up to 136 weeks
Incidence and severity of TEAEs in patients treated with cemiplimab in combination with other agents | Up to 136 weeks
Incidence and severity of TEAEs in patients treated with fianlimab in combination with cemiplimab without chemotherapy | Up to 136 weeks
Incidence and severity of TEAEs in patients treated with fianlimab in combination with cemiplimab with chemotherapy | Up to 136 weeks
PK of cemiplimab: Cmax | Up to 136 weeks
  Peak serum concentration
PK of cemiplimab: tmax | Up to 136 weeks
  Time to Cmax
PK of cemiplimab: Ctrough | Up to 136 weeks
  Drug concentration in serum at the end of a dosing interval
PK of cemiplimab: Area under the drug concentration-time curve in serum (AUC3w) | Up to 136 weeks
  AUC over a 3-week dosing interval
PK of cemiplimab: t½ estimated over a 3-week dosing interval | Up to 136 weeks
  Observed terminal half-life

SECONDARY OUTCOMES:
Immunogenicity against cemiplimab and fianlimab | Up to 136 weeks
  Evaluate the immunogenicity of cemiplimab and fianlimab after single-dose administration
Objective Response Rate (ORR) | Up to 135 weeks
  As assessed by an Independent Review Committee (IRC) using RECIST 1.1 (Eisenhauer 2009) in Part 2, Cohorts A and C
Duration of Response (DOR) | Up to 136 weeks
  As assessed by an IRC (per RECIST1.1) in Part 2, Cohorts A and C

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (20):
- Japan (20):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Kurume University Hospital, Kurume, Fukuoka
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Kanagawa Cancer Center - Thora, Yokohama, Kanagawa
  - Sasebo City General Hospital, Sasebo, Nagasaki
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Kansai Medical University Hirakata Hospital, Hirakata, Osaka
  - Osaka Metropolitan University Hospital, Osaka, Osaka
  - National Hospital Organization Kinki-chuo Chest Medical Center, Sakai-shi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka
  - Saitama Cancer Center, Shinden, Saitama
  - National Cancer Center Hospital - Tsukiji Campus, Chuo Ku, Tokyo
  - Hiroshima City Hiroshima Citiz, Hiroshima
  - Nagasaki University Hospital, Nagasaki
  - Osaka International Cancer Institute, Osaka
  - Tokushima University Hospital, Tokushima

REFERENCES:
- [Derived] Kitano S, Shimizu T, Koyama T, Ebata T, Iwasa S, Kondo S, Shimomura A, Fujiwara Y, Yamamoto N, Paccaly A, Li S, Rietschel P, Sims T. Dose exploration results from Phase 1 study of cemiplimab, a human monoclonal programmed death (PD)-1 antibody, in Japanese patients with advanced malignancies. Cancer Chemother Pharmacol. 2021 Jan;87(1):53-64. doi: 10.1007/s00280-020-04161-6. Epub 2020 Nov 4. PMID 33146741